CLINICAL TRIAL: NCT05669989
Title: International, Multi-center, Open-label, Treatment Extension Study in Patients With Multiple Myeloma Who Are Still Benefitting From Isatuximab-based Therapy Following Completion of a Phase 1, 2, or 3 Parental Study
Brief Title: International Treatment-extension Study in Adult Participants With Multiple Myeloma and Who Have Derived Clinical Benefit From Isatuximab
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS17704; U1111-1277-6635 (Registry Identifier: ICTRP); 2023-507180-19 (Registry Identifier: CTIS); 2022-002253-26 (EudraCT Number)
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; cemiplimab; Dexamethasone; Lenalidomide; pomalidomide; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Isatuximab (Experimental): Participants will receive isatuximab as monotherapy or in a combination regimen, according to the treatment the participant received on the parental protocol
  Interventions: Drug: Isatuximab intravenous (IV); Drug: Cemiplimab (SAR439684); Drug: Dexamethasone; Drug: Lenalidomide; Drug: Pomalidomide; Drug: Isatuximab subcutaneous (SC); Drug: Carfilzomib

INTERVENTIONS:
Drug: Isatuximab intravenous (IV) — Route of administration: IV infusion; Pharmaceutical form: Vial
  Other Names: SARCLISA®, SAR650984
Drug: Cemiplimab (SAR439684) — Route of administration: IV infusion; Pharmaceutical form: Vial
Drug: Dexamethasone — Route of administration: Oral or IV infusion; Pharmaceutical form: Tablets/single use vial
Drug: Lenalidomide — Route of administration: Oral; Pharmaceutical form: Capsules
Drug: Pomalidomide — Route of administration: Oral; Pharmaceutical form: Hard capsules
Drug: Isatuximab subcutaneous (SC) — Route of administration: SC injection with the investigational isatuximab injector device; Pharmaceutical form: Vial
  Other Names: SARCLISA®, SAR650984
Drug: Carfilzomib — Route of administration: IV infusion; Pharmaceutical form: Vial

SUMMARY:
* This is a multi-center, open-label, Phase 2 treatment extension study in participants with multiple myeloma who are still benefitting from isatuximab based therapy following completion of a Phase 1, 2, or 3 parental study.
* This Treatment Extension study has the purpose to provide continued access to isatuximab. Adult participants with multiple myeloma who have enrolled on an isatuximab parental study for which study objectives are completed will be eligible to be enrolled in this Treatment Extension study.
* The primary objective of the study is to assess long-term safety of isatuximab as study treatment.

DETAILED DESCRIPTION:
Participants can continue the treatment until disease progression, unacceptable adverse events, participant wish to discontinue study treatment, study treatment is commercially available and reimbursed in participant's country, or for any other reason, whichever comes first. The overall study duration will be of approximately 42 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years of age (or the legal age of consent in the jurisdiction in which the study is taking place), at the time of signing the informed consent.
* Participants of a parental Phase 1, 2, or 3 clinical study assessing isatuximab monotherapy or in a combination regimen with all the study objectives completed.
* Participants still receiving isatuximab at the time of the parental study closure, who are continuing to benefit from isatuximab as monotherapy or in combination, as determined by the treating physician, and who meet the criteria to initiate a subsequent cycle of therapy as described in the parental study protocol. A participant not receiving isatuximab at the end of the parental study who does not have access locally to the ongoing treatment may also be included.
* Contraception (with double contraception methods) for male and female participants; not pregnant or breastfeeding for female participants; no sperm donation for male participants.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Participant has evidence of progressive disease during or at the time of the parental study closure.
* Participant has not recovered to ≤Grade 2 from nonhematologic AEs (as per NCI CTCAE v5.0) related to any anticancer therapy received prior to signing informed consent on the extension study.
* As the latest line of treatment participant received an antimyeloma therapy other than the isatuximab-based therapy in the parental study before the first IMP in this study.
* Individuals accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalized.
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.
* Participants are employees of the clinical study site or other individuals directly involved in the conduct of the study, or immediate family members of such individuals.
* Any country-related specific regulation that would prevent the participant from entering the study.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events | Baseline to 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (37):
- Washington University- Site Number : 8400001, St Louis, Missouri, United States
- Australia (6):
  - Investigational Site Number : 0360006, Blacktown, New South Wales
  - Investigational Site Number : 0360001, Saint Leonards, New South Wales
  - Investigational Site Number : 0360003, Wollongong, New South Wales
  - Investigational Site Number : 0360004, Melbourne, Victoria
  - Investigational Site Number : 0360005, Melbourne, Victoria
  - Investigational Site Number : 0360002, Richmond, Victoria
- Brazil (3):
  - Hospital Mae de Deus- Site Number : 0760003, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo - HCFMUSP- Site Number : 0760002, São Paulo, São Paulo
  - Instituto Americas - Ensino, Pesquisa e Inovação - Rio de Janeiro - Avenida Jorge Curi- Site Number : 0760001, Rio de Janeiro
- Investigational Site Number : 1520001, Temuco, Chile
- Investigational Site Number : 1560001, Tianjin, China
- Czechia (3):
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2030003, Ostrava
  - Investigational Site Number : 2030001, Prague
- Investigational Site Number : 2460001, Helsinki, Finland
- Investigational Site Number : 2500002, Nantes, France
- Greece (3):
  - Investigational Site Number : 3000004, Athens
  - Investigational Site Number : 3000003, Athens
  - Investigational Site Number : 3000001, Pátrai
- Investigational Site Number : 3800002, Torino, Italy
- Investigational Site Number : 3920001, Okayama, Japan
- New Zealand (2):
  - Investigational Site Number : 5540002, Auckland
  - Investigational Site Number : 5540001, Wellington
- Russia (2):
  - Investigational Site Number : 6430002, Kirov
  - Investigational Site Number : 6430001, Moscow
- South Korea (2):
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
- Spain (7):
  - Investigational Site Number : 7240006, Seville, Andalusia
  - Investigational Site Number : 7240004, Santander, Cantabria
  - Investigational Site Number : 7240005, Badalona, Catalunya [Cataluña]
  - Investigational Site Number : 7241001, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240001, Pamplona, Navarre
  - Investigational Site Number : 7240003, Madrid
  - Investigational Site Number : 7240002, Salamanca
- Investigational Site Number : 7520004, Luleå, Sweden
- Investigational Site Number : 1580001, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org